CLINICAL TRIAL: NCT05628597
Title: Effects of the Fos Biomedical Device on Diabetes Risk Factors and Sleep Quality in Adults at Risk for Type 2 Diabetes: A Randomized, Placebo-controlled, Crossover Trial
Brief Title: Effects of Fos Biomedical Device on Diabetes Risk Factors and Sleep Quality in Adults at Risk for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Griffin Hospital (Other)
Collaborators: Fos Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021-10
Record Dates: First submitted 2021-10-14; First posted 2022-11-28 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Pre Diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: To provide a sound basis for the statistical comparison of outcome measures for treatment assignments, participants will be randomized to 1 of 2 sequence permutations of the Fos Biomedical patch product and a placebo patch product, which will begin after randomization. Each permutation will include a 12-week treatment phase, followed by a 2-month washout phase, followed by a 12-week treatment phase (8 months total for each study participant, including the washout phase).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigators and study participants will be blinded to treatment assignments. Each of the two patch products (Fos Biomedical product and placebo) will be provided to the study team by the study funder (Fos Biomedical). The products will have a similar appearance and texture. One will be described to study participants and study team members as "Product A" and the other as "Product B." The description of products A and B will be sent by Fos Biomedical in a sealed envelope that will be kept in locked cabinet at the PRC. The envelope will be opened at the conclusion of the statistical analyses. Therefore all members of the investigative team will be blinded to the study interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fos Biomedical patch product (Active Comparator): Participants will be randomized to 1 of 2 sequence permutations of the Fos Biomedical patch product and a placebo patch product, which will begin after randomization.
  Interventions: Device: Fos Biomedical patch product; Device: Fos Biomedical patch product:placebo
- Fos Biomedical product: placebo (Placebo Comparator): Participants will be randomized to 1 of 2 sequence permutations of the Fos Biomedical patch product and a placebo patch product, which will begin after randomization.
  Interventions: Device: Fos Biomedical patch product; Device: Fos Biomedical patch product:placebo

INTERVENTIONS:
Device: Fos Biomedical patch product — Participants will apply a Fos Biomedical patch system (consisting of 2 single-use patches) on a daily basis for 12 weeks.
Device: Fos Biomedical patch product:placebo — Participants will apply a placebo patch system (consisting of 2 single-use patches) on a daily basis for 12 weeks.

SUMMARY:
Purpose Phototherapy has an array of potential benefits in human health. The effects of a non-transdermal Fos Biomedical product (which utilizes the concept of phototherapy) on diabetes risk factors and sleep quality in people at risk for type 2 diabetes are unclear. Proposed is a single-blind randomized crossover placebo-controlled trial to assess the impact of daily use of the Fos Biomedical product for a 12-week period on cardio-metabolic risk factors and self-reported sleep quality among adults at risk for type 2 diabetes.

Specific Aims

* To determine the effects of the use of the Fos Biomedical product daily for 12 weeks, as compared to placebo patch, on glycemic control in adults at risk for type 2 diabetes. Specifically, to show that the use of the Fos Biomedical product for 12 weeks, as compared to placebo patch, will improve glycated hemoglobin in adults at risk for type 2 diabetes.
* To assess the effects of the use of the Fos Biomedical product, versus placebo patch, for a 12-week period on insulin sensitivity, serum lipids, C-reactive protein, anthropometric measures, self-reported sleep quality, and endothelial function in adults at risk for type 2 diabetes. Specifically, to show clinically meaningful improvement or neutral effects in insulin sensitivity, serum lipids, C-reactive protein, anthropometric measures, self-reported sleep quality, and endothelial function in adults at risk for type 2 diabetes.
* To assess the impact of Fos Biomedical product on liver function and kidney function in adults at risk for type 2 diabetes

Hypotheses

* Daily use of the Fos Biomedical product for 12 weeks will improve glycated hemoglobin in adults at risk for type 2 diabetes.
* Daily use of the Fos Biomedical product for 12 weeks will improve or have neutral effects on insulin sensitivity, serum lipids, C-reactive protein, anthropometric measures, self-reported sleep quality and endothelial function in adults at risk for type 2 diabetes.
* The use of the Fos Biomedical product will have no clinically meaningful adverse effects on liver function and kidney function in adults at risk for type 2 diabetes.

DETAILED DESCRIPTION:
Background Pre-diabetes is a serious medical condition associated with elevated blood glucose that is higher than normal, but not high enough to be considered for a diagnosis of diabetes. An estimated 88 million adults aged 18 years and older have pre-diabetes in the United States (U.S.), yet more than 84% of those with pre-diabetes are unaware. Those with pre-diabetes are at increased risk for developing diabetes, cardiovascular disease (CVD), and stroke. Fifteen to 30% of individuals with pre-diabetes are likely to develop type 2 diabetes mellitus (T2DM) within 5 years. Pre-diabetes is a major risk factor associated with metabolic syndrome. Insulin resistance and excess body weight are common in both pre-diabetes and metabolic syndrome.

Metabolic syndrome - a cluster of risk factors that increase the risk of T2DM and CVD - affects about 35% of adults in the U.S. The risk factors for metabolic syndrome include hypertension, dyslipidemia, hyperglycemia, and excess body weight (especially due to excess central body fat). These risk factors represent an independent risk for developing T2DM, CVD, and stroke, as well as an increased risk of mortality. The risk of T2DM, CVD, and stroke increases with the number of metabolic risk factors. Persons with metabolic syndrome, when compared with healthy persons, have a 5-fold increased risk for T2DM. The combination of pre-diabetes and metabolic syndrome compared with healthy persons is associated with an even higher (i.e., 21-fold) risk for T2DM.

An inconsistent sleep schedule or a general lack of sleep has been associated with increased risk of developing T2DM. Specifically, sleep disturbance is associated with pre-diabetes and metabolic syndrome. Sleep disturbance is associated with poor cardio-metabolic control (i.e., hypertension, dyslipidemia, and a reduction in insulin level released after eating). Further, elevated stress hormones that keep the body awake have been associated with increased blood glucose level by increasing the production of glucose in the liver; decreasing glucose uptake in the muscles and fat cells; decreasing insulin secretion; and increasing insulin resistance. In addition, sleep deprivation has also been associated with increased appetite, which heightens the risk of T2DM. Again, insufficient sleep has been associated with higher levels of ghrelin, which increase appetite, and lower levels of leptin, which signals fullness. Therefore, improving sleep patterns has the potential to improve cardio-metabolic risk factors among those at risk for T2DM.

Lifestyle practices that promote good sleep hygiene and reduce stress have been associated with lower risk of T2DM and the control of cardio-metabolic risk factors among those at risk for T2DM. In addition, consistent sleep patterns have also been associated with improved glycemic control in T2DM. Phototherapy is thought to help improve sleep patterns in persons with circadian rhythm sleep disorders to normal sleeping patterns and times. Further, in a meta-analysis phototherapy therapy was shown to improve symptoms of vascular complications and quality of life that are linked to diabetes. In animal models, phototherapy has been shown to reduce abdominal fat. In addition, phototherapy has also been associated with improved insulin sensitivity in T2DM.

Phototherapy, also known as photobiomodulation (PBM), or low-level light therapy, has been known for almost 50 years but still has not gained widespread acceptance, largely due to uncertainty about the mechanisms of action. In recent years, much knowledge has been gained in this area. The primary site of light absorption in mammalian cells has been identified as the mitochondria, and more specifically, cytochrome c oxidase (CCO), an enzyme that contains both heme and copper centers and is known to reduce oxygen to water at the end of the mitochondrial respiratory chain. CCO has recently been shown to have an additional enzymatic activity: the reduction of nitrite to nitric oxide (NO) upon exposure to low-intensity light. The absorption peaks of CCO are in the visible (420-450 nm and 600-700 nm) and the near-infrared (760-980 nm) spectral region.

The leading hypothesis is that photons dissociate inhibitory NO from CCO, leading to an increase in electron transport, mitochondrial membrane potential and ATP production. Another hypothesis concerns light-sensitive ion channels that can be activated, allowing calcium to enter the cell. After the initial photon absorption events, numerous signaling pathways are activated via reactive oxygen species (ROS), cyclic AMP, NO and Ca2+, leading to activation of transcription factors. These transcription factors can lead to increased expression of genes related to protein synthesis, cell migration and proliferation, anti-inflammatory signaling, anti-apoptotic proteins, and antioxidant enzymes.

In a recent study showing that PBM reduced blood glucose and insulin resistance and reversed metabolic abnormalities in skeletal muscle in two diabetic mouse models, PBMT accelerated adenosine triphosphate (ATP) and ROS generation by elevating CCO activity. ROS-induced activation of phosphatase and tensin homolog (PTEN)/ protein kinase B (AKT) signaling after PBMT promoted glucose transporter GLUT4 translocation and glycogen synthase activation, accelerating glucose uptake and glycogen synthesis in skeletal muscle.

The effects of the non-transdermal Fos Biomedical patch system (which utilizes the concept of phototherapy) on cardio-metabolic risk factors and sleep quality in persons at risk for T2DM are unclear. Proposed is a randomized crossover placebo-controlled trial to assess the impact of the Fos Biomedical patch system use on cardio-metabolic risk factors and sleep quality among adults at risk for type 2 diabetes. Specifically, the investigators hypothesize that the use of the Fos Biomedical patch system for 12 weeks, as compared to placebo patch system, will improve glycated hemoglobin, other markers of cardio-metabolic risk factors and sleep quality in adults at risk for T2DM.

ELIGIBILITY:
Inclusion Criteria:

(1) Males > 40 years of age; (2) Post-menopausal females not currently on hormone replacement therapy; (3) Non-smokers; (4) Overweight with BMI ≥25kg/m²; (5) At risk for type 2 diabetes as defined by meeting at least one of the criteria listed below: (i) Metabolic syndrome, i.e. meet three out of five of the following criteria:

1. Blood pressure >130/85 mmHg or currently taking antihypertensive medication;
2. Fasting plasma glucose (FPG) >100 mg/dL (6.1 mmol/L);
3. Serum triglycerides level (TG)>150 mg/dL (1.69 mmol/L);
4. High-density lipoprotein (HDL) cholesterol level < 40 mg/dL (1.04 mmol/L) in men, and < 50 mg/dL (1.29 mmol/L) in women;
5. Waist circumference of >40 inches (102 cm) for men and > 35 inches (88 cm) for women; fasting blood glucose >100mg/dL and <126mg/dL.

(ii) Hemoglobin A1C in the range of 5.7-6.4%

Exclusion Criteria:

1. Failure to meet inclusion criteria;
2. Anticipated inability to complete study protocol for any reason;
3. Type 1 or type 2 diabetes;
4. Personal history or family history of skin cancer;
5. Having lupus;
6. Having liver disease;
7. Use of lipid-lowering or antihypertensive medications, unless stable on medication for at least 3 months and willing to refrain from taking medication for 12 hours prior to clinical outcome measures assessment;
8. Regular use of high doses of vitamin E or C;
9. Use of insulin, glucose-sensitizing medication, vasoactive medication (including glucocorticoids, antineoplastic agents, psychoactive agents, or bronchodilators) or nutraceuticals;
10. Regular use of fiber supplements;
11. Sleep apnea;
12. Coagulopathy, known bleeding diathesis, or history of clinically significant hemorrhage; or current use of warfarin.
13. Known allergic or dermatological reactions to any of the components of the patch product or placebo - polyethylene, silicone, or acrylate adhesive - that could have contact with the skin of study participants during their use of the product.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin | Baseline, 12 weeks, 20 weeks, 32 weeks
  Glycated hemoglobin (HbA1c) will be measured to assess the average concentration. HbA1c predicts the average amount of plasma glucose. The study team will use HbA1c to gauge the average amount of blood glucose level over a previous 3-month period.

SECONDARY OUTCOMES:
Insulin sensitivity | Baseline, 12 weeks, 20 weeks, 32 weeks
  Glucose and insulin will be measured at each time point. Participants will be asked to fast at least 8 hours before glucose and insulin measurement. Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) will be calculated based on the fasting glucose and insulin levels to gauge the impact of phototherapy on glycemic control in the study participants. HOMA-IR will be calculated according to the formula: fasting insulin (µU/mL) multiplied by fasting glucose (mg/dL) divided by 405.
Percent body fat | Baseline, 12 weeks, 20 weeks, 32 weeks
  Percent body fat will be measured on the Tanita SC-240 Body Composition Analyzer using bioelectrical impedance analysis, which uses the resistance of electrical flow through the body to estimate body fat.
Visceral fat rating | Baseline, 12 weeks, 20 weeks, 32 weeks
  Visceral fat rating will be measured on the Tanita SC-240 Body Composition Analyzer.
Total body water percent | Baseline, 12 weeks, 20 weeks, 32 weeks
  Total water body water percent will be measured on the Tanita SC-240 Body Composition Analyzer.
Body weight | Baseline, 12 weeks, 20 weeks, 32 weeks
  Body weight will be measured for all study participants during each visit. It will be measured to the nearest 0.5 pound using a balance-type medical scale. Subjects will be measured in the morning (fasting), unclothed with the exception of undergarments.
Body mass index (BMI) | Baseline, 12 weeks, 20 weeks, 32 weeks
  Body mass index (BMI) will be measured as a participant's weight in kilograms divided by the participant's height in meters squared.
Waist circumference | Baseline, 12 weeks, 20 weeks, 32 weeks
  Waist circumference will be measured using the U.S. government standard protocol. It will be measured around the narrowest point between ribs and hips when viewed from the front after exhaling.
Office blood pressure (BP) | Baseline, 12 weeks, 20 weeks, 32 weeks
  Systolic and diastolic BP will be measured at each visit using an approved automated device. Blood pressure will be measured (average of two measurements, with five minutes between measurements) with the participant sitting in a quiet room.
C-reactive protein (CRP) | Baseline, 12 weeks, 20 weeks, 32 weeks
  Serum CRP values will be determined using a high sensitivity CRP (hsCRP) ELISA method.
Serum lipids | Baseline, 12 weeks, 20 weeks, 32 weeks
  Total cholesterol (Tchol), triglycerides (TG), and high-density lipoprotein (HDL) will be obtained by direct measurements. Very-low-density lipoprotein (VLDL) and low-density-lipoprotein (LDL) will be obtained by calculation: VLDL = TG/5; and LDL = Tchol - (VLDL + HDL). HDL:Tchol ratio will be used to evaluate the impact of treatment assignments on the lipid panel
Endothelial function (EF) | Baseline, 12 weeks, 20 weeks, 32 weeks
  The brachial artery reactivity studies (BARS) methodology to be employed is as described in the published "Guidelines for Ultrasound Assessment of Endothelial-dependent Flow-mediated Vasodilation of the Brachial Artery." The measure of interest is flow-mediated dilatation (FMD) of the brachial artery.
Dietary pattern | Baseline, 12 weeks, 20 weeks, 32 weeks
  To assess differences in diet quality and help the study team track any variation in dietary pattern over the course of the study, participants will be asked at baseline, 6 weeks and 12 weeks to provide information on the foods and beverages that they consumed during a 3-day period (i.e., 2 weekdays and 1 weekend day). For each 3-day period, participants will complete 3 consecutive 24-hour recalls using a web-based Automated Self-Administered 24-Hour Recall (ASA24) (available from the National Cancer Institute at http://riskfactor.cancer.gov/tools/instruments/asa24/), which will guide them through the process of completing the recall data, and these data will be reviewed by the study dietitian.
Physical activity | Baseline, 12 weeks, 20 weeks, 32 weeks
  Physical activity will be determined by the Seven-Day Physical Activity Recall [PAR]. 41 The PAR is one of the most widely used physical activity assessments in exercise science and epidemiological research. The popularity of this measure stems largely from its versatility and relative ease of use for research applications. The PAR provides detail regarding the duration, intensity, and volume (energy expenditure) of physical activity and can therefore be used for a variety of applications. Because it utilizes a one-week time frame, the data from the PAR is often considered representative of typical activity patterns. While it requires considerable cognitive effort by the participants, the interviewer-administered version can be completed in a reasonable amount of time (~20 minutes).
Pittsburgh Sleep Quality Index (PSQI) | Baseline, 12 weeks, 20 weeks, 32 weeks
  The PSQI questionnaire will be used to assess the self-reported quality of participants' sleep before and after each intervention phase. The PSQI is a self-rated questionnaire to assess perceived sleep quality and disturbances over a 1-month time interval. This 19-item instrument uses a Likert scale (ranging from 0 to 3) to assess seven clinically derived domains of sleep: sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. Clinical and clinimetric properties of the PSQI were assessed over an 18-month period with "good" vs. "poor" sleepers. A global score > 5 yielded a diagnostic sensitivity of 89.6% and specificity of 86.5% (kappa = 0.75, p < 0.001) in distinguishing good vs. poor sleepers.
Liver function | Baseline, 12 weeks, 20 weeks, 32 weeks
  Liver function will be assessed based on serum levels of aspartate transaminase (AST) and alanine aminotransferase (ALT).
Kidney function | Baseline, 12 weeks, 20 weeks, 32 weeks
  Kidney function will be assessed based on serum creatinine levels.
Medication use | Baseline, 12 weeks, 20 weeks, 32 weeks
  The study team will track any changes in medication use.
Compliance | Baseline, 12 weeks, 20 weeks, 32 weeks
  For each of the two treatment assignment periods, good compliance will be defined as >80% use of treatment during the respective 12-week treatment assignment. During the study assessment visit at the end of each treatment assignment, the study coordinator will meet with participants to assess compliance to the treatment assignment. Compliance will be assessed by self-report and by collecting the returned product use log at the end of each 12-week treatment assignment.

CONTACTS AND LOCATIONS:
Overall Officials: Valentine Y Njike, MD, MPH, Principal Investigator — Yale-Griffin Prevention Research Center
Locations (1):
- Yale-Griffin Prevention Research Center, Derby, Connecticut, United States

REFERENCES:
- [Derived] Njike VY, Ayettey RG, Treu JA, Comerford BP, Onuigbo M. Cardio-metabolic health and sleep quality in adults at risk for Type 2 Diabetes using the Fos Biomedical Non-Transdermal Patch System via photo-biomodulation: A randomized, placebo-controlled crossover trial. Contemp Clin Trials Commun. 2025 Feb 15;44:101448. doi: 10.1016/j.conctc.2025.101448. eCollection 2025 Apr. PMID 40115254